CLINICAL TRIAL: NCT02342860
Title: Measuring the Impact of WASH in Schools in the Lao People's Democratic Republic
Brief Title: The Impact of Improved WASH in Schools on Absence, Diarrhea and Helminth Infection in Lao PDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: UNICEF (Other)
Responsible Party: Principal Investigator, Matthew Freeman, MPH, PhD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00076404
Record Dates: First submitted 2015-01-09; First posted 2015-01-21 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Hygiene
Keywords: Water; sanitation; hygiene access in school
MeSH Terms: interventions — Therapeutic Irrigation; Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WASH in Schools (WinS) programme (Experimental): Schools in the intervention group will receive the UNICEF/Department of Foreign Affairs and Trade (DFAT)-supported WinS programme that includes a new water supply, 3 latrines (boys, girls, handicapped), and handwashing facilities. It will also include behavior change education.
  Interventions: Other: WASH in Schools (WinS) programme
- Control (No Intervention): Schools in the control group will receive no additional WinS programming.

INTERVENTIONS:
Other: WASH in Schools (WinS) programme — The intervention group will receive the UNICEF/DFAT-supported WinS programme, which consists of the following intervention package:
  * Hardware: water supply system, handwashing station for group handwashing, and gender-segregated toilets with one facility accessible to students with physical disabilities;
  * Software: operations and maintenance (O&M) training for teachers, hygiene training, and basic hygiene package.
  Arms: WASH in Schools (WinS) programme

SUMMARY:
The investigators will conduct a cluster-randomized trial to assess the impact of a school-based water, sanitation and hygiene program on health and educational outcomes of school children in Saravane Province, Laos. The intervention will include an improved water supply (borehole), a sanitation block that includes three pour-flush latrines with rainwater harvesting to be used for flushing and a urinal, and sinks for handwashing with soap. The school will also receive a facility for group handwashing (large pipe where many children can wash hands at once. United Nations International Children's Emergency Fund (UNICEF) will additionally provide behavior change education. Our key outcome of interest is pupil absence, which will be measured longitudinally using roll-call on days of schools visits. Secondary outcomes include self-reported absence, diarrhea and respiratory infection of a random selection of students. The investigators will also monitor the fidelity of the intervention and assess school conditions and pupil sanitation and handwashing behaviors using structured observation.

DETAILED DESCRIPTION:
Though limited, research suggests school-based water, sanitation and hygiene (WASH) improvements are capable of reducing pupil absence from 35-42%. However, few studies have rigorously evaluated the impact of comprehensive WASH in Schools (WinS) improvements on pupil absenteeism; to date, no research on the impact of WinS has been conducted in Lao PDR. This study will use longitudinal data collection to quantify the impact of UNICEF's WinS program on pupil learning and health in Lao People's Democratic Republic (Lao PDR).

Research activities will take place Saravane Province, Lao PDR. Schools are eligible if they are a primary, non-Community-Built Construction (CBC) school, and lacking WASH facilities. A total of 136 schools will be randomly selected from a pool of all eligible schools, and randomly assigned to either the intervention or comparison group (68 schools each). Directors of the selected schools will be contacted and informed about procedures prior to the start of the study, and they will provide permission to conduct the study at their schools if they so choose. At each school the investigators will randomly select up to 60 pupils in grades 1-5. Research staff will approach selected pupils at school to request informed oral assent for participation. The informed assent process and data collection will be conducted by local trained enumerators in the child's preferred language of Laotian or a local dialect. Oral rather than written assent was chosen due to varied literacy capabilities and to limit paperwork that identifies participants. A waiver of parental consent for pupil interviews has been secured from the Ministry of Education and Sports. At each school, school directors will be asked to sign in loco parentis ("in the place of parent") on behalf of the pupil participants.

Data collection will take place at each school once every six to eight weeks for the duration of up to three school years. The investigators will conduct school observations and an interview with the school director about school conditions, handwashing behavior observations of children, and a review of aggregate school-wide academic record data including percentage of children obtaining a passing average, advancing to the next class, and drop-outs. None of these school activities collect personal data or identifiers. Data collection with pupils will be done with the same pupils every six to eight weeks and will entail a five-minute interview asking about recent absence, symptoms of diarrhea or respiratory illness, age, and grade. Select pupils in a subset of schools will undergo testing for cognition, attention, and hydration. Select pupils in a subset of school will provide a stool sample for analyses of helminth infection prior to school-wide de-worming. Data collection will also take place at the household of select pupils in a subset of schools. The investigators will conduct a household survey once at the beginning of each school year to assess the range of household WASH access among pupils in study selected schools.

All data collection will occur at the school or the household, will be conducted by trained local enumerators, and will be stored on password-protected mobile data collection devices. Data will be uploaded to a password-protected server and will not contain personal identifying information, but rather a pupil identification . Enumerators will maintain a separate form that links identifications with names of pupils, which will be kept confidential. There are no direct benefits other than contribution to general knowledge that will inform future school WASH projects. There are no risks to participation other than a small amount of class time missed by pupils, and great efforts will be made to minimize time outside of class.

ELIGIBILITY:
Schools must meet the following criteria to be eligible for inclusion in the study:

* Located in the Saravane, Ta Oy, Toumlane, Lakhonepheng, Vapy, Khongsedone, Lao Ngam, and Samoui Districts
* Non-Community-Based Construction (CBC) school
* Primary school
* Lacking functional WASH facilities
* If part of a complex, no other schools in the complex have already been selected to participate in the study.

Pupils must meet the following criteria to be eligible for inclusion in the study:

* Grades 3-5 in study selected schools
* Understand and respond to study assent process

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8873 (Actual)
Dates: Start 2014-09; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Pupil absenteeism | 20 months
  Rates of pupil absenteeism from school, measured through roll call, review of teacher records, and pupil self-report

SECONDARY OUTCOMES:
Pupil educational attainment ( measured through review of school/teacher records) | 20 months
  Enrollment, attrition, progression, and performance will be measured through review of school/teacher records
Pupil health attainment (measured through pupil self-report) | 20 months
  Diarrhea, respiratory infection, and conjunctivitis will be measured through pupil self-report; hydration will be measured through analysis of urine specific gravity; helminth prevalence and infection intensity will be measured through analysis of stool samples
Behavior change (Handwashing behavior and proxy indicators of WASH facility usage will be measured using structured observation) | 20 months
  Handwashing behavior and proxy indicators of WASH facility usage will be measured using structured observation; household and school WASH facility usage will be measured through pupil self-report

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Freeman, PhD, MPH, Principal Investigator — Emory University

REFERENCES:
- [Result] Chard AN, Freeman MC. Design, Intervention Fidelity, and Behavioral Outcomes of a School-Based Water, Sanitation, and Hygiene Cluster-Randomized Trial in Laos. Int J Environ Res Public Health. 2018 Mar 22;15(4):570. doi: 10.3390/ijerph15040570. PMID 29565302
- [Derived] Chard AN, Levy K, Baker KK, Tsai K, Chang HH, Thongpaseuth V, Sistrunk JR, Freeman MC. Environmental and spatial determinants of enteric pathogen infection in rural Lao People's Democratic Republic: A cross-sectional study. PLoS Negl Trop Dis. 2020 Apr 8;14(4):e0008180. doi: 10.1371/journal.pntd.0008180. eCollection 2020 Apr. PMID 32267881